CLINICAL TRIAL: NCT04018508
Title: Pilot Study of Massage Therapy to Improve Self-efficacy in Patients With Left-ventricular Device
Brief Title: Massage Therapy for Self-efficacy in LVAD Recipients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID19 pandemic closed in-person clinics; LVAD surgeon left institution, stopping LVAD implants
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Hunter Groninger, Investigator, Medstar Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00000591; NCT04851236 (obsolete NCT alias)
Record Dates: First submitted 2019-06-13; First posted 2019-07-12 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure
Keywords: left ventricular assist device; massage; coping; self efficacy
MeSH Terms: conditions — Heart Failure | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massages (Experimental): During routine clinic visits, subjects will receive a total of six 30-minute massages (one massage per week for 4 weeks, then one massage every two weeks for 4 weeks).
  Interventions: Other: Massage
- Control (No Intervention): Subjects randomized to the control arm will also attend routine clinic visits at the same pre-prescribed intervals (one clinic visit per for 4 weeks, then one visit every two weeks for 4 weeks).

INTERVENTIONS:
Other: Massage — Massage intervention including effleurage, petrissage and energy work/Reiki at a pressure of 2 or less (Walton Pressure Scale)
  Arms: Massages

SUMMARY:
This pilot study evaluates the role of massage therapy to improve self-efficacy in patients with advanced heart failure who have recently received a left-ventricular assist device. In addition to usual care, half of the volunteer patients will receive a massage at regular clinic visits and half will not receive any massage.

DETAILED DESCRIPTION:
Patients with advanced heart failure who undergo left-ventricular assist device (LVAD) implantation may experience notable physical and/or emotional distress associated with this lifestyle-changing procedure. Furthermore, these patients are faced with the task of coping with the trauma of surgery, creating new self-care routines, and learning to live with a lifesaving mechanical device that must always be connected to a power source.The immediate weeks and months after LVAD implantation are a critical period to lower physical and emotional distress and to influence patient coping and adaptation. In small studies, massage therapy has been increasingly used to improve patient self-efficacy and coping. In this pilot study, we investigate whether regularly scheduled massages delivered in the clinic setting improve self-efficacy and coping in this select patient population.

ELIGIBILITY:
Inclusion Criteria:

* capacitated, at least 18 years of age, received LVAD implant during last hospital admission

Exclusion Criteria:

* incapacitated, non-English speaking, negative pressure isolation, unstable spine, very low serum platelets (<10,000/uL), received massage in 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Change in Self-Efficacy for Managing Chronic Disease 6-item Scale from Baseline to Repeat Visits | 1) Baseline; 2) after week 4; 3) after week 8; 4) 1 month post completion
  The Self-Efficacy for Managing Chronic Disease 6-item Scale is a psychometric scale that asks the subject 6 questions regarding confidence managing aspects of the chronic illness (fatigue, physical discomfort, emotional distress, non-pain symptoms, medication adherence, completing assigned health care related tasks). Subjects respond to each question on a Likert scale from zero to 10 (zero="not confident at all"; 10="totally confident"). The score for the scale is the mean of the composite scores of the 6 Likert scales.

SECONDARY OUTCOMES:
Change in score on Brief COPE Inventory from baseline to repeat visits | 1) Baseline; 2) after week 4; 3) after week 8; 4) 1 month post completion
  The Brief COPE is a 28-item multidimensional measure of strategies used for coping or regulating cognitions in response to stressors. This abbreviated inventory (based on the complete 60-item COPE Inventory) is comprised of items that assess the frequency with which a person uses different coping strategies (e.g., "I've been turning to work or other activities to take my mind off things," "I've been making fun of the situation," "I've been criticizing myself") rated on a scale from 1, I haven't been doing this at all, to 4, I've been doing this a lot. There are 14 two-item subscales within the Brief COPE, and each is analyzed separately: (1) self-distraction, (2) active coping, (3) denial, (4) substance use, (5) use of emotional support, (6) use of instrumental support, (7) behavioral disengagement, (8) venting, (9) positive reframing, (10) planning, (11) humor, (12) acceptance, (13) religion, and (14) self-blame.
Change in score on National Comprehensive Cancer Network Distress Thermometer from baseline to repeat visits | 1) Baseline; 2) after week 4; 3) after week 8; 4) 1 month post completion
  The NCCN Distress Thermometer asks the patient to report his/her distress on a scale between 0 (no distress) and 10 (extreme distress). The number provided on the scale is the patient's score.
Change in score on McGill Quality of Life Scale (Revised) from baseline to repeat visits | 1) Baseline; 2) after week 4; 3) after week 8; 4) 1 month post completion
  The McGill Quality of Life Questionnaire (Revised) is a 15-item multidimensional tool designed to measure physical well-being, physical symptoms, psychological symptoms, existential well-being and support, as well as overall quality of life. Created for people at all stages of a life-threatening illness (from diagnosis to cure or death), the MQOL(Revised) was designed to assess general domains applicable to all clients/patients, incorporate the existential domain, balance physical and nonphysical aspects of quality of life, and include both positive and negative influences on quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No